CLINICAL TRIAL: NCT06219590
Title: Acetylcholine Iontophoresis As A New Challenge With Type 2 Diabetic Peripheral Neuropathy: A Possible New Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Reham Abdelrazek Mohamed Ellisy, Principal investigator., South Valley University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ach Iontophoresis neuropathy
Record Dates: First submitted 2023-10-27; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes Mellitus; Peripheral Neuropathy
Keywords: Acetylcholine iontophoresis; diabetic neuropathy; electrophysiological investigations; Nitric oxide; type2 diabetes mellitus; aerobic exercises
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Peripheral Nervous System Diseases; Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (A) (Active Comparator): * 40 patients with type 2 diabetes mellitus clinically proved peripheral neuropathy.
  * Both groups were received conventional medical treatment and healthy diet.
  * Group A was received iontophoresis by acetylcholine with (15) min for three sessions per week for four weeks.
  Interventions: Procedure: Acetylcholine Iontophoresis
- Control group (B) (Sham Comparator): * 40 patients with asymptomatic type 2 diabetes mellitus, both groups were selected from south valley university hospitals.
  * Both groups were received conventional medical treatment and healthy diet.
  * Group (B) was received shame iontophoresis with (15) min for three sessions per week for four weeks.
  Interventions: Procedure: Shame Acetylcholine Iontophoresis

INTERVENTIONS:
Procedure: Acetylcholine Iontophoresis — Acetylcholine Iontophoresis 15 min/ three sessions/ week for two weeks.
  Arms: Study group (A)
Procedure: Shame Acetylcholine Iontophoresis — Shame Acetylcholine Iontophoresis 15 min/ three sessions/ week for two weeks.
  Arms: Control group (B)

SUMMARY:
The investigators initial study opened the way for randomized trials that monitor the effects of acetylcholine (Ach) iontophoresis vasodilators on endothelial nitric oxide synthetase (NOS) to develop a transdermal treatment that is effective, free from systemic adverse effects.

DETAILED DESCRIPTION:
The investigators studied endothelial-mediated microvascular blood flow in neuropathic diabetic patients to determine the association between endothelial regulation of the microcirculation and the expression of endothelial constitutive nitric oxide synthetase (NOS). As a result, the nerve fibers can become damaged. Once the nerves have been damaged they cannot repair themselves.

Material and methods:

A group of 80 patients (male and female) diagnosed as type 2 diabetes mellitus, will be included in the study their age ranged from 40-60 years. Patients randomly will be divided into two groups:

Study groups (A) 40 patients type 2 diabetes mellitus with clinically proved peripheral neuropathy. And control group (B) 40 patients with asymptomatic type 2 diabetes mellitus. They were selected from south valley university hospitals. Group (A) receive iontophoresis by acetylcholine with (15) min for three sessions per week for four weeks. Also the investigators followed up study group (A) one month of aerobic exercises in form of 15 minute walking, bicycling, or swimming, and the investigators reevaluated nitric oxide level. Group (B) received shame iontophoresis with (15) min for three sessions per week for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients have to be symptomatically stable with type 2 diabetes mellitus complicated with peripheral neuropathy.
* Optimized pharmacological treatment that will be remained unchanged throughout the study.

Exclusion Criteria:

* Implanted cardiac pacemakers.
* Patients with known skin allergies.
* Presence of skin inflammations.
* Peripheral vascular disease.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-28 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Role of acetylcholine iontophoresis in improving Nitric oxide level in diabetic peripheral neuropathy patients. | one month (baseline assessment and after one month of Ach iontophoresis and exercise)
  Blood samples were withdrawn from visible peripheral veins by venipuncture then centrifuged and serum was used for nitric oxide level assessment (No micromole/liter) , Nitric oxide measured using commercially available calorimetric assay kits using spectrophotometer (chem7 erba, labomed, Germany). Suspected improvement in nitric oxide level by acetylcholine iontophoresis, patient will receive three sessions iontophoresis weekly for one month and No will be assessed baseline and post assay will be done pre (baseline) and post acetylcholine iontophoresis exposure and aerobic exercise.
Electrophysiological assessment of patients with acetylcholine iontophoresis and Ach iontophoresis role in improving diabetic peripheral neuropathy | one month (baseline assessment and after one month of Ach iontophoresis and exercise)
  Nerve conduction velocity of nerves and needle EMG of upper limb and lower limbs will be assessed pre and post exposure, expecting improvement in nerve conduction velocity (expressed latency ms, amplitude mv).
Numerical rating pain scale | One month
  Patient just say the level of pain feeling, zero means no pain, while 10 means most intense pain possible. Expecting pain improvement after one month of Ach iontophoresis and exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, South Valley University, Qina, Egypt

REFERENCES:
- [Background] Abularrage CJ, Sidawy AN, Aidinian G, Singh N, Weiswasser JM, Arora S. Evaluation of the microcirculation in vascular disease. J Vasc Surg. 2005 Sep;42(3):574-81. doi: 10.1016/j.jvs.2005.05.019. PMID 16171612
- [Background] Alzahrani SH, Ajjan RA. Coagulation and fibrinolysis in diabetes. Diab Vasc Dis Res. 2010 Oct;7(4):260-73. doi: 10.1177/1479164110383723. Epub 2010 Sep 16. PMID 20847109
- [Background] Goyal M, Kumar A, Mahajan N, Moitra M. 2013: Treatment of plantar fasciitis by taping vs. iontophoresis: a randomized clinical trial. J Exercise Sci Physiother; 9:34-39.
- [Background] Barwick AL, Tessier JW, Janse de Jonge X, Ivers JR, Chuter VH. Peripheral sensory neuropathy is associated with altered postocclusive reactive hyperemia in the diabetic foot. BMJ Open Diabetes Res Care. 2016 Jul 7;4(1):e000235. doi: 10.1136/bmjdrc-2016-000235. eCollection 2016. PMID 27486520